CLINICAL TRIAL: NCT06023498
Title: Optimizing Impact of Manual Therapy and Exercise on Lumbar Spinal Stenosis With Neurogenic Claudication: A Multi-Site Feasibility Study
Brief Title: Optimizing Impact of Manual Therapy on Lumbar Spinal Stenosis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Boston Medical Center (Other); VA Pittsburgh Healthcare System (U.S. Federal Agency); Syracuse VA Medical Center (U.S. Federal Agency); Orlando VA Medical Center (U.S. Federal Agency); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Debra Weiner, Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY24010020; R01AT012534 (NIH)
Record Dates: First submitted 2023-08-14; First posted 2023-09-05 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-08

CONDITIONS: Lumbar Spinal Stenosis
MeSH Terms: conditions — Spinal Stenosis | interventions — Musculoskeletal Manipulations; Exercise

STUDY DESIGN:
Intervention Model Description: Randomized controlled clinical trial - feasibility study
Who Masked: Outcomes Assessor
Masking Description: Performance-based outcomes measures will be collected by a research coordinator who is masked to participant group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Manual Therapy and Exercise (MTE) (Experimental): Participants will be asked to attend 10 sessions of manual therapy that will be administered by a chiropractic physician and will consist of movements designed to enhance flexibility and muscle health. Session will last ~ 20 minutes.
  The home exercise program (HEP) will consist of a light aerobic program (either walking with the lumbar spine in slight flexion while supported by a wheeled walker, going up and down a flight of stairs, using a treadmill, or using an exercise bicycle), neural mobilization self-stretches, individualized muscular stretches and core strengthening exercises. Participants will be encouraged to do the HEP 1-2 times per day, starting with 5 minutes and working up to 30 minutes.
  During the subsequent 6 months, there will be no additional treatment administered. Participants will be asked to continue their HEP.
  Interventions: Other: Manual Therapy and Exercise
- MTE Plus MTE Boosters (Experimental): Participants will be asked to attend 10 sessions of manual therapy that will be administered by a chiropractic physician and will consist of movements designed to enhance flexibility and muscle health. Session will last ~ 20 minutes.
  The home exercise program (HEP) will consist of a light aerobic program (either walking with the lumbar spine in slight flexion while supported by a wheeled walker, going up and down a flight of stairs, using a treadmill, or using an exercise bicycle), neural mobilization self-stretches, individualized muscular stretches and core strengthening exercises. Participants will be encouraged to do the HEP 1-2 times per day, starting with 5 minutes and working up to 30 minutes.
  During the subsequent 6 months, participants will be asked to return for monthly MTE booster sessions, and they will be asked to continue their HEP.
  Interventions: Other: Manual Therapy and Exercise
- MTE and Intramuscular Electroacupuncture (IMEA) Plus MTE and IM Boosters (Experimental): Participants will be asked to attend 10 sessions of manual therapy that will be administered by a chiropractic physician and will consist of movements designed to enhance flexibility and muscle health. Session will last ~ 20 minutes.
  Participants also will be asked to attend weekly intramuscular electroacupuncture (IMEA) sessions administered by a licensed acupuncturist. 30-gauge acupuncture needles will be placed in the muscles of the lower back and buttocks and gentle pulsing electrical stimulation will be delivered for 20 minutes.
  The home exercise program (HEP) will be identical to that in the MTE and the MTE + Boosters groups.
  During the subsequent 6 months, participants will be asked to return for monthly MTE and IMEA boosters. Participants also will be asked to continue their HEP.
  Interventions: Other: Manual Therapy and Exercise; Other: Intramuscular Electroacupuncture

INTERVENTIONS:
Other: Manual Therapy and Exercise — The 20-minute manual therapy procedures will include:
  * Distraction-manipulation: manually assisted segmental lumbar traction manipulation using a specialized treatment table
  * Neural mobilization: rhythmic stretches of the sciatic and femoral nerves75
  * Hip, sacroiliac and lumbar facet mobilizations to improve joint mobility
  * Soft tissue mobilization of lumbopelvic and lower extremity muscles using manual pressure over taut bands/myofascial trigger points and post-isometric (contract-relax) stretching techniques.
Other: Intramuscular Electroacupuncture — As described previously
  Arms: MTE and Intramuscular Electroacupuncture (IMEA) Plus MTE and IM Boosters

SUMMARY:
Lumbar spinal stenosis, a common condition in older adults, can cause pain and difficulty walking (i.e., intermittent neurogenic claudication - INC). Patients with INC not infrequently undergo spinal surgery that fails to help them 1/3-1/2 the time. The purpose of this multi-site feasibility study is to prepare for the conduct of a randomized controlled trial to test the efficacy of manual therapy, exercise, and intramuscular electroacupuncture in reducing pain and improving walking ability for those with INC, and ultimately limiting the need for surgical referrals.

DETAILED DESCRIPTION:
Decompressive laminectomy (DL), the most common spinal surgery in older adults, is performed to alleviate lumbar spinal stenosis (LSS) and reduce associated pain, paresthesias, and/or weakness when walking (i.e., intermittent neurogenic claudication - INC). The PI's recent prospective cohort study of 193 older veterans followed for 12 months following DL revealed that over 50% of participants did not experience significant functional improvement. Similar rates of failed surgery have been reported in non-veteran populations. Since the vast majority of DLs are performed electively, non-surgical treatment is recommended as an initial step. Two clinical trials have demonstrated modest efficacy of manual therapy and exercise (MTE) for people with INC that was sustained in one trial, but not in the other. Recent clinical practice guidelines recommend adding acupuncture as a non-surgical pain management strategy and highlight the need for high quality evidence to support this recommendation. The investigators' clinical experience and preliminary research data regarding the efficacy of electroacupuncture (specifically, intramuscular electroacupuncture [IMEA]) in these patients are promising. Ultimately, the study team wishes to conduct a randomized controlled clinical trial to optimize and sustain the efficacy of MTE by potentially a) increasing the robustness of the initial response via addition of IMEA and b) its durability via boosters. This two-site feasibility study will be conducted at Boston Medical Center and the Orlando VA Medical Center, chosen because of their sociodemographic diversity and prevalence of patients with multiple comorbidities, characteristics that will ultimately facilitate broad generalizability of study findings. The study team will evaluate the feasibility of recruiting, randomizing and retaining participants; fidelity of intervention delivery; participant adherence to prescribed interventions; and the accuracy and completeness of data collection procedures. Sixty participants (30 per site) with imaging-identified LSS and INC who have not had lumbar surgery, will be randomized to receive 1) MTE for 3 months (10 sessions over 12 weeks) followed by a 6-months observation period; 2) MTE for 3 months followed by monthly MTE booster sessions for 6-months; OR 3) MTE + IMEA for 3 months followed by monthly MTE + IMEA for 6-months. The primary outcome (Brigham Spinal Stenosis questionnaire) for the future efficacy trial will be measured at baseline, 3 months (primary endpoint), 6 and 9 months. The study also will measure community mobility (life space), emotional functioning (PHQ8 and GAD7), pain medications, and other key parameters relevant to older adults with LSS and INC (e.g., smoking, BMI, medical comorbidity). Fidelity will be optimized by delivering standardized provider training, conducting regular review of participant provider intervention sessions and documentation, and monthly all-site huddles. The study also will monitor participant attendance and home exercise compliance. If the study demonstrates feasibility (primary outcome for this study) of the proposed methods, the study team will be positioned to test a new model of care for patients with LSS and INC designed to optimize their function and quality of life and save substantial morbidity and healthcare resources.

ELIGIBILITY:
Inclusion Criteria:

* Intermittent neurogenic claudication (INC), defined as pain or discomfort with walking or prolonged standing that radiates beyond the spinal area and is relieved with sitting (ascertained using a structured interview)

  * Average pain/discomfort severity > moderate
  * Advanced imaging (e.g., MRI, CT scan, CT-myelogram) evidence of lumbar spinal stenosis (extracted from electronic medical record, or outside report provided by participant; advanced imaging will not be performed as part of our study procedures)
  * Able to commit to 9 months of study participation
  * English speaking

Exclusion Criteria:

* Red flags indicative of serious underlying illness requiring urgent care (e.g., fever, change in bowel/ bladder function, sudden severe change in pain, unintentional weight loss, new leg weakness)
* Walking capacity over 2 miles
* Other conditions that significantly impact mobility (e.g., painful conditions such as advanced hip/knee osteoarthritis with pain more severe than INC pain, Parkinson's disease, stroke, vascular claudication, angina pectoris, pulmonary disease, morbid obesity (i.e., BMI > 40).
* Prior lumbar surgery, because of its negative impact on spinal biomechanics;
* Positive screen for dementia (i.e., Folstein Mini-Mental State Examination);
* Acute medical or psychiatric illness, or active substance abuse that renders the patient incapable of being a reliable study participant;
* Prohibitive communication impairment (e.g., severe hearing or visual impairment)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-06-11 (Actual); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants recruited and retained after 9 months of participation | Number of participants recruited at each of two study sites over a period of 12 months (duration of recruitment period) - assessed at 12 months after recruitment starts; number of participants retained at each site after 9 months of study participation
  Number of participants recruited and retained at each site
Median number of intervention sessions attended | 3 months (at completion of initial intervention) and 9 months (at completion of follow up period)
  Median number of intervention sessions attended at each site
Rate of missing data | Baseline, 3 months, and 9 months
  Percentage of study data that are not entered into data collection system

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Orlando VA Medical Center, Orlando, Florida
  - Boston Medical Center, Boston, Massachusetts

DOCUMENTS (1):
  • Informed Consent Form (2025-01-14): https://cdn.clinicaltrials.gov/large-docs/98/NCT06023498/ICF_000.pdf